CLINICAL TRIAL: NCT04715932
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study of Hesperidin Therapy on COVID-19 Symptoms: The Hesperidin Coronavirus Study (Hesperidin)
Brief Title: Study of Hesperidin Therapy on COVID-19 Symptoms (HESPERIDIN)
Acronym: Hesperidin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Ingenew Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHICC-2020-003
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Anosmia; Fever; Cough; Shortness of Breath; Sore Throat; Nausea; Vomiting; Headache; Muscle Weakness; Pain, Muscle; Pain, Chest; Pain, Joint; Pain, Abdominal; Pain; Irritable Mood; Confusion
MeSH Terms: conditions — COVID-19; Anosmia; Fever; Cough; Dyspnea; Pharyngitis; Nausea; Vomiting; Headache; Muscle Weakness; Myalgia; Chest Pain; Arthralgia; Abdominal Pain; Pain; Confusion | interventions — Hesperidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hesperidin 1000mg (Active Comparator): Patients will receive study medication Hesperidin and will take 2 capsules of 500mg at the same time in the evening, at bedtime with water.
  Interventions: Drug: Hesperidin
- Placebo 1000mg (Placebo Comparator): Patients will receive study medication Placebo and will take 2 capsules of 500mg at the same time in the evening, at bedtime with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hesperidin — Patients will receive study medication Hesperidin and will take 2 capsules of 500mg at the same time in the evening, at bedtime with water.
  Arms: Hesperidin 1000mg
Drug: Placebo — Patients will receive study medication Placebo and will take 2 capsules of 500mg at the same time in the evening, at bedtime with water.
  Arms: Placebo 1000mg

SUMMARY:
The main aim of this study is to determine the effects of short-term treatment with hesperidin on COVID-19 symptoms in comparison with a placebo. Treatment effects will be observed through a symptoms diary that will be completed by participants throughout the study and by taking the oral temperature daily.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled study. The study will include subjects from Quebec diagnosed with COVID-19 infections. Following informed consent, 216 subjects meeting all inclusion and no exclusion criteria will be randomized to receive either hesperidin 1000 mg once daily (q.d.)) or placebo (1:1 allocation ratio) for 14 days. Investigational drug will be delivered to the patients' homes with an electronic oral thermometer and a symptoms diary. Follow-up phone assessments will occur after 3, 7, 10, and 14 days following randomization for evaluation of COVID-19 symptoms. Electronic Case Report Form (eCRF) will be completed by the research personnel over the phone with the patients. The symptoms diary will be mailed back to the coordinating center at the end of the study in a pre-addressed envelope.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 positive by polymerase chain reaction (PCR) testing;
* Participant must be able to evaluate their symptoms and report them in the symptoms diary;
* Patients must be able to take their oral temperature daily with an electronic thermometer provided to them with study materials;
* Males and females, at least 18 years of age, capable and willing to provide informed consent;
* Female patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing at least one method of contraception and preferably two complementary forms of contraception including a barrier method (e.g. male or female condoms, spermicides, sponges, foams, jellies, diaphragm, intrauterine device (IUD)) throughout the study;
* Patient must have received a diagnosis of COVID-19 infection within the last 48 hours and have one or more symptoms;
* Outpatient setting (not currently hospitalized or under immediate consideration for hospitalization);
* Patient must be able and willing to comply with the requirements of this study protocol.

Exclusion Criteria:

* Patient currently hospitalized or under immediate consideration for hospitalization;
* Patient currently in shock or with hemodynamic instability;
* Patient undergoing chemotherapy for cancer;
* Patient is unable to take oral temperature using an electronic thermometer;
* Patient who received at least one dose of the COVID-19 vaccine;
* Female patient who is pregnant or breast-feeding or is considering becoming pregnant during the study;
* People taking anticoagulant/antiplatelet medications, those with bleeding disorders, and people two weeks before or after surgery;
* Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study;
* Regular consumption of natural products containing more than 150 mg of hesperidin or regular consumption of more than 1 glass of orange juice per day;
* Known allergy to any of the medicinal and non-medicinal ingredient: hesperidin, microcrystalline cellulose, magnesium stearate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Dupuis, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 216 subjects were randomized into the study with 109 assigned to placebo and 107 to hesperidin.
Period: Overall Study
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Started | 107 | 109
Completed | 106 | 109
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hesperidin 1000mg | Placebo 1000mg | Total
Number analyzed (Participants) | 107 | 109 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.31 (13.02) | 40.67 (11.26) | 40.98 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 119
  Male | 48 | 49 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 104 | 105 | 209
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 102 | 107 | 209
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: KG/m^2] | 28.12 (6.38) | 28.21 (6.82) | 28.16 (6.59)
Diabetes [Count of Participants; unit: Participants]
  With Diabetes | 6 | 1 | 7
  Without Diabetes | 101 | 108 | 209
Hypertension [Count of Participants; unit: Participants]
  With Hypertension | 14 | 9 | 23
  Without Hypertension | 93 | 100 | 193
Respiratory Disease [Count of Participants; unit: Participants]
  With Respiratory Disease | 15 | 18 | 33
  Without Respiratory Disease | 92 | 91 | 183
Asthma [Count of Participants; unit: Participants]
  With Asthma | 14 | 17 | 31
  Without Asthma | 93 | 92 | 185
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants]
  With COPD | 0 | 1 | 1
  Without COPD | 107 | 108 | 215
Pulmonary Fibrosis [Count of Participants; unit: Participants]
  With Pulmonary Fibrosis | 1 | 0 | 1
  Without Pulmonary Fibrosis | 106 | 109 | 215
Other Respiratory Disease [Count of Participants; unit: Participants]
  With Other Respiratory Disease | 0 | 1 | 1
  Without Other Respiratory Disease | 107 | 108 | 215

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With COVID-19 Symptoms at Day 3.
Description: Number of subjects with any of the following COVID-19 symptoms: fever (temperature > 38 degrees), cough, shortness of breath or anosmia, at day 3.
Time Frame: Day 3
Population: Number of patients analysed differs from the number of patients assigned to the arm or comparison group as not all subjects replied to the questionnaire or follow-up call, whether a symptom occurred or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  Subject has at least one of the selected COVID-19 symptoms. | 93 | 90
  Subject has none of the selected COVID-19 symptoms. | 9 | 13
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.3849, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.60 to 3.69]

2. Primary Outcome: Number of Subjects With COVID-19 Symptoms at Day 7.
Description: Number of subjects with any of the following COVID-19 symptoms: fever (temperature > 38 degrees), cough, shortness of breath or anosmia, at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 101
Participants
  Subject has at least one of the selected COVID-19 symptoms. | 74 | 76
  Subject has none of the selected COVID-19 symptoms. | 17 | 25
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.3139, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.71 to 2.88]

3. Primary Outcome: Number of Subjects With COVID-19 Symptoms at Day 10.
Description: Number of subjects with any of the following COVID-19 symptoms: fever (temperature > 38 degrees), cough, shortness of breath or anosmia, at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 99
Participants
  Subject has at least one of the selected COVID-19 symptoms. | 58 | 60
  Subject has none of the selected COVID-19 symptoms. | 32 | 39
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5886, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.65 to 2.14]

4. Primary Outcome: Number of Subjects With COVID-19 Symptoms at Day 14.
Description: Number of subjects with any of the following COVID-19 symptoms: fever (temperature > 38 degrees), cough, shortness of breath or anosmia, at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 94
Participants
  Subject has at least one of the selected COVID-19 symptoms. | 39 | 55
  Subject has none of the selected COVID-19 symptoms. | 40 | 39
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.2328, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.38 to 1.27]

5. Secondary Outcome: Mean Number of COVID-19 Symptoms at Day 3.
Description: Mean number of COVID-19 symptoms (range 0-13) at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Symptoms
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 101 | 102
Symptoms | 4.74 (2.52) | 4.16 (2.39)
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.1560, Mixed Models Analysis; Generalized linear mixed model (repeated poisson regression); Rate Ratio = 1.14, 95% CI 2-sided [0.95 to 1.37]

6. Secondary Outcome: Mean Number of COVID-19 Symptoms at Day 7.
Description: Mean number of COVID-19 symptoms (range 0-13) at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Symptoms
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 101
Symptoms | 3.13 (2.49) | 2.96 (2.46)
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.6233, Mixed Models Analysis; Generalized linear mixed model (repeated poisson regression); Rate Ratio = 1.06, 95% CI 2-sided [0.84 to 1.33]

7. Secondary Outcome: Mean Number of COVID-19 Symptoms at Day 10.
Description: Mean number of COVID-19 symptoms (range 0-13) at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Symptoms
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 99
Symptoms | 2.01 (2.19) | 1.95 (2.12)
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8290, Mixed Models Analysis; Generalized linear mixed model (repeated poisson regression); Rate Ratio = 1.03, 95% CI 2-sided [0.78 to 1.37]

8. Secondary Outcome: Mean Number of COVID-19 Symptoms at Day 14.
Description: Mean number of COVID-19 symptoms (range 0-13) at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Symptoms
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 94
Symptoms | 1.38 (1.76) | 1.40 (1.65)
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.9222, Mixed Models Analysis; Generalized linear mixed model (repeated poisson regression); Rate Ratio = 0.98, 95% CI 2-sided [0.69 to 1.40]

9. Secondary Outcome: Number of Subjects With Complete Disappearance of Any Symptom.
Description: The descriptive statistics are the number of participants having complete disappearance of any symptom.
Time Frame: From randomization to occurence of first event, assessed up to 14 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 106 | 106
Participants
  Complete disappearance of COVID-19 symptoms after randomization | 29 | 33
  No complete disappearance of COVID-19 symptoms after randomization | 77 | 73
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8834, Log Rank

10. Secondary Outcome: Number of Subjects With the Cough Symptom.
Description: Number of subjects with the cough symptom at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With Cough Symptom | 54 | 54
  Without Cough Symptom | 48 | 49
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.9416, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.59 to 1.77]

11. Secondary Outcome: Number of Subjects With the Cough Symptom.
Description: Number of subjects with the cough symptom at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With Cough Symptom | 37 | 45
  Without Cough Symptom | 54 | 57
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.6296, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.49 to 1.55]

12. Secondary Outcome: Number of Subjects With the Cough Symptom.
Description: Number of subjects with the cough symptom at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With Cough Symptom | 26 | 35
  Without Cough Symptom | 64 | 65
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.3711, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.41 to 1.40]

13. Secondary Outcome: Number of Subjects With the Cough Symptom.
Description: Number of subjects with the cough symptom at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With Cough Symptom | 21 | 29
  Without Cough Symptom | 58 | 66
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5696, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.42 to 1.61]

14. Secondary Outcome: Number of Subjects With the Presence of Fever.
Description: Number of subjects with the presence of fever (temperature > 38 degrees) at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 101 | 102
Participants
  With the presence of fever | 5 | 6
  Without the presence of fever | 96 | 96
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.7583, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.26 to 2.67]

15. Secondary Outcome: Number of Subjects With the Presence of Fever.
Description: Number of subjects with the presence of fever (temperature > 38 degrees) at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 101
Participants
  With the presence of fever | 3 | 4
  Without the presence of fever | 87 | 97
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8091, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.20 to 3.58]

16. Secondary Outcome: Number of Subjects With the Presence of Fever.
Description: Number of subjects with the presence of fever (temperature > 38 degrees) at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 99
Participants
  With the Presence of Fever | 3 | 2
  Without the Presence of Fever | 87 | 97
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5591, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.30 to 9.42]

17. Secondary Outcome: Number of Subjects With the Presence of Fever.
Description: Number of subjects with the presence of fever (temperature > 38 degrees) at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 94
Participants
  With the presence of fever | 0 | 1
  Without the presence of fever | 79 | 93
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.9983, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression)

18. Secondary Outcome: Number of Subjects With the Presence of Shortness of Breath.
Description: Number of subjects with the presence of shortness of breath at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of shortness of breath | 46 | 35
  Without the presence of shortness of breath | 56 | 68
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.1068, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.90 to 2.82]

19. Secondary Outcome: Number of Subjects With the Presence of Shortness of Breath.
Description: Number of subjects with the presence of shortness of breath at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of shortness of breath | 28 | 30
  Without the presence of shortness of breath | 63 | 72
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8382, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.57 to 1.98]

20. Secondary Outcome: Number of Subjects With the Presence of Shortness of Breath.
Description: Number of subjects with the presence of shortness of breath at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of shortness of breath | 19 | 18
  Without the presence of shortness of breath | 71 | 82
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5912, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.59 to 2.51]

21. Secondary Outcome: Number of Subjects With the Presence of Shortness of Breath.
Description: Number of subjects with the presence of shortness of breath at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of shortness of breath | 14 | 13
  Without the presence of shortness of breath | 65 | 82

22. Secondary Outcome: Number of Subjects With the Presence of Anosmia.
Description: Number of subjects with the presence of anosmia at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of anosmia | 52 | 59
  Without the presence of anosmia | 50 | 44
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.3686, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.45 to 1.35]

23. Secondary Outcome: Number of Subjects With the Presence of Anosmia.
Description: Number of subjects with the presence of anosmia at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of anosmia | 43 | 47
  Without the presence of anosmia | 48 | 55
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8711, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.59 to 1.86]

24. Secondary Outcome: Number of Subjects With the Presence of Anosmia.
Description: Number of subjects with the presence of anosmia at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of anosmia | 34 | 37
  Without the presence of anosmia | 56 | 63
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.9124, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.57 to 1.87]

25. Secondary Outcome: Number of Subjects With the Presence of Anosmia.
Description: Number of subjects with the presence of anosmia at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of anosmia | 20 | 31
  Without the presence of anosmia | 59 | 64
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.2952, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.36 to 1.37]

26. Secondary Outcome: Number of Subjects With the Presence of Feverish or Chills.
Description: Number of subjects with the presence of feverish or chills at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of feverish or chills | 24 | 21
  Without the presence of feverish or chills | 78 | 82
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5894, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.62 to 2.34]

27. Secondary Outcome: Number of Subjects With the Presence of Feverish or Chills.
Description: Number of subjects with the presence of feverish or chills at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of feverish or chills | 10 | 10
  Without the presence of feverish or chills | 81 | 92
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.7887, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.45 to 2.89]

28. Secondary Outcome: Number of Subjects With the Presence of Feverish or Chills.
Description: Number of subjects with the presence of feverish or chills at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of feverish or chills | 4 | 6
  Without the presence of feverish or chills | 86 | 94
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.6348, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.20 to 2.70]

29. Secondary Outcome: Number of Subjects With the Presence of Feverish or Chills.
Description: Number of subjects with the presence of feverish or chills at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of feverish or chills | 1 | 3
  Without the presence of feverish or chills | 78 | 92
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.4257, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.04 to 3.92]

30. Secondary Outcome: Number of Subjects With the Presence of Sore Throat.
Description: Number of subjects with the presence of sore throat at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of sore throat | 33 | 23
  Without the presence of sore throat | 69 | 80
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.1113, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.89 to 3.11]

31. Secondary Outcome: Number of Subjects With the Presence of Sore Throat.
Description: Number of subjects with the presence of sore throat at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of sore throat | 17 | 13
  Without the presence of sore throat | 74 | 89
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.2613, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.71 to 3.47]

32. Secondary Outcome: Number of Subjects With the Presence of Sore Throat.
Description: Number of subjects with the presence of sore throat at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of sore throat | 6 | 8
  Without the presence of sore throat | 84 | 92
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.7273, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.27 to 2.49]

33. Secondary Outcome: Number of Subjects With the Presence of Sore Throat.
Description: Number of subjects with the presence of sore throat at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of sore throat | 3 | 4
  Without the presence of sore throat | 76 | 91
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8909, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.19 to 4.19]

34. Secondary Outcome: Number of Subjects With the Presence of Runny Nose.
Description: Number of subjects with the presence of runny nose at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of runny nose | 48 | 38
  Without the presence of runny nose | 54 | 65
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.1438, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.87 to 2.67]

35. Secondary Outcome: Number of Subjects With the Presence of Runny Nose.
Description: Number of subjects with the presence of runny nose at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of runny nose | 25 | 22
  Without the presence of runny nose | 66 | 80
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.3440, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.71 to 2.68]

36. Secondary Outcome: Number of Subjects With the Presence of Runny Nose.
Description: Number of subjects with the presence of runny nose at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of runny nose | 18 | 17
  Without the presence of runny nose | 72 | 83
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5968, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.58 to 2.56]

37. Secondary Outcome: Number of Subjects With the Presence of Runny Nose.
Description: Number of subjects with the presence of runny nose at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of runny nose | 12 | 10
  Without the presence of runny nose | 67 | 85
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.3620, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.62 to 3.76]

38. Secondary Outcome: Number of Subjects With the Presence of Nausea/Vomiting.
Description: Number of subjects with the presence of nausea/vomiting at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of nausea/vomiting | 21 | 12
  Without the presence of nausea/vomiting | 81 | 91
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.0875, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.91 to 4.27]

39. Secondary Outcome: Number of Subjects With the Presence of Nausea/Vomiting.
Description: Number of subjects with the presence of nausea/vomiting at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of nausea/vomiting | 9 | 11
  Without the presence of nausea/vomiting | 82 | 91
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8397, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.36 to 2.32]

40. Secondary Outcome: Number of Subjects With the Presence of Nausea/Vomiting.
Description: Number of subjects with the presence of nausea/vomiting at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of nausea/vomiting | 6 | 5
  Without the presence of nausea/vomiting | 84 | 95
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.6265, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.40 to 4.65]

41. Secondary Outcome: Number of Subjects With the Presence of Nausea/Vomiting.
Description: Number of subjects with the presence of nausea/vomiting at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of nausea/vomiting | 2 | 2
  Without the presence of nausea/vomiting | 77 | 93
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8528, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.16 to 8.91]

42. Secondary Outcome: Number of Subjects With the Presence of Headache.
Description: Number of subjects with the presence of headache at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of headache | 48 | 41
  Without the presence of headache | 54 | 62
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.2983, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.77 to 2.35]

43. Secondary Outcome: Number of Subjects With the Presence of Headache.
Description: Number of subjects with the presence of headache at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of headache | 34 | 34
  Without the presence of headache | 57 | 68
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5611, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.66 to 2.16]

44. Secondary Outcome: Number of Subjects With the Presence of Headache.
Description: Number of subjects with the presence of headache at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of headache | 22 | 20
  Without the presence of headache | 68 | 80
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.4643, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.65 to 2.58]

45. Secondary Outcome: Number of Subjects With the Presence of Headache.
Description: Number of subjects with the presence of headache at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of headache | 10 | 9
  Without the presence of headache | 69 | 86
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5063, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.53 to 3.62]

46. Secondary Outcome: Number of Subjects With the Presence of General Weakness.
Description: Number of subjects with the presence of general weakness at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of general weakness | 63 | 55
  Without the presence of general weakness | 39 | 48
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.2292, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.80 to 2.47]

47. Secondary Outcome: Number of Subjects With the Presence of General Weakness.
Description: Number of subjects with the presence of general weakness at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of general weakness | 39 | 40
  Without the presence of general weakness | 52 | 62
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.6097, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.65 to 2.07]

48. Secondary Outcome: Number of Subjects With the Presence of General Weakness.
Description: Number of subjects with the presence of general weakness at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of general weakness | 20 | 21
  Without the presence of general weakness | 70 | 79
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8389, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.54 to 2.16]

49. Secondary Outcome: Number of Subjects With the Presence of General Weakness.
Description: Number of subjects with the presence of general weakness at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of general weakness | 14 | 17
  Without the presence of general weakness | 65 | 78
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.9764, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.45 to 2.17]

50. Secondary Outcome: Number of Subjects With the Presence of Pain.
Description: Number of subjects with the presence of pain at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of pain | 44 | 50
  Without the presence of pain | 58 | 53
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.4403, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.46 to 1.40]

51. Secondary Outcome: Number of Subjects With the Presence of Pain.
Description: Number of subjects with the presence of pain at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of pain | 17 | 23
  Without the presence of pain | 74 | 79
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.5112, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.39 to 1.60]

52. Secondary Outcome: Number of Subjects With the Presence of Pain.
Description: Number of subjects with the presence of pain at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of pain | 13 | 14
  Without the presence of pain | 77 | 86
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.9306, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.46 to 2.36]

53. Secondary Outcome: Number of Subjects With the Presence of Pain.
Description: Number of subjects with the presence of pain at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of pain | 5 | 8
  Without the presence of pain | 74 | 87
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.6046, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.23 to 2.36]

54. Secondary Outcome: Number of Subjects With the Presence of Irritability/Confusion.
Description: Number of subjects with the presence of irritability/confusion at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of irritability/confusion | 20 | 18
  Without the presence of irritability/confusion | 82 | 85
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.6963, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.57 to 2.34]

55. Secondary Outcome: Number of Subjects With the Presence of Irritability/Confusion.
Description: Number of subjects with the presence of irritability/confusion at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of irritability/confusion | 6 | 10
  Without the presence of irritability/confusion | 85 | 92
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.4250, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.22 to 1.88]

56. Secondary Outcome: Number of Subjects With the Presence of Irritability/Confusion.
Description: Number of subjects with the presence of irritability/confusion at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of irritability/confusion | 4 | 4
  Without the presence of irritability/confusion | 86 | 96
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8797, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.27 to 4.65]

57. Secondary Outcome: Number of Subjects With the Presence of Irritability/Confusion.
Description: Number of subjects with the presence of irritability/confusion at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of irritability/confusion | 3 | 1
  Without the presence of irritability/confusion | 76 | 94
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.2634, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 3.71, 95% CI 2-sided [0.37 to 37.03]

58. Secondary Outcome: Number of Subjects With the Presence of Diarrhea.
Description: Number of subjects with the presence of diarrhea at day 3.
Time Frame: Day 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 102 | 103
Participants
  With the presence of diarrhea | 22 | 16
  Without the presence of diarrhea | 80 | 87
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.2710, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.73 to 3.06]

59. Secondary Outcome: Number of Subjects With the Presence of Diarrhea.
Description: Number of subjects with the presence of diarrhea at day 7.
Time Frame: Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 91 | 102
Participants
  With the presence of diarrhea | 15 | 10
  Without the presence of diarrhea | 76 | 92
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.1748, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.77 to 4.30]

60. Secondary Outcome: Number of Subjects With the Presence of Diarrhea.
Description: Number of subjects with the presence of diarrhea at day 10.
Time Frame: Day 10
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 90 | 100
Participants
  With the presence of diarrhea | 6 | 6
  Without the presence of diarrhea | 84 | 94
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.8513, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.34 to 3.63]

61. Secondary Outcome: Number of Subjects With the Presence of Diarrhea.
Description: Number of subjects with the presence of diarrhea at day 14.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
Number analyzed (Participants) | 79 | 95
Participants
  With the presence of diarrhea | 4 | 4
  Without the presence of diarrhea | 75 | 91
Statistical Analysis 1: Comparison: Hesperidin 1000mg vs Placebo 1000mg; Test type: Superiority; p = 0.7906, Mixed Models Analysis; Generalized linear mixed model (repeated binary logistic regression); Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.29 to 5.07]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between randomization/baseline until the end of study visit (up to 14 days).
Description: Subjects reporting multiple TEAEs within a given system organ class/preferred term were counted only once within the category.
  Results are based on safety population. Table of adverse events includes serious adverse events. Number of Participants at Risk differs from the number of participants assigned to the arm or comparison group. One participant from the placebo group is not part of the safety population. However, "All-Cause Mortality" is on the intention to treat population.
Arm/Group | Hesperidin 1000mg | Placebo 1000mg
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/109
Serious Adverse Events (participants affected / at risk) | 4/107 | 1/108
Other Adverse Events (participants affected / at risk) | 20/107 | 16/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hesperidin 1000mg (N=107) | Placebo 1000mg (N=108)
Arthritis bacterial (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hesperidin 1000mg (N=107) | Placebo 1000mg (N=108)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 4
Pneumonia (Infections and infestations) | 4 | 3
Sinusitis (Infections and infestations) | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Only one dosage regimen of hesperidin was tested in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT04715932/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT04715932/SAP_001.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT04715932/ICF_002.pdf